CLINICAL TRIAL: NCT06304961
Title: A Randomised, Single-dose, Parallel Group Study in Healthy Volunteers to Assess the Relative Bioavailability of Two Different Dosage Forms for Tozorakimab Via Subcutaneous Administration
Brief Title: A Study to Investigate Relative Bioavailability of Two Different Dosage Forms for Tozorakimab Via Subcutaneous Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9180C00011
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy Participants
Keywords: Human immunoglobulin G1 monoclonal antibody; Chronic Obstructive Pulmonary Disease; Asthma; Pharmacokinetics; Bioavailability
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tozorakimab Dosage form A (Test) (Experimental): Participants will receive a single dose of Tozorakimab Dosage form A via subcutaneous (SC) injection.
  Interventions: Biological: Tozorakimab
- Tozorakimab Dosage form B (Reference) (Experimental): Participants will receive a single dose of Tozorakimab Dosage form B via SC injection.
  Interventions: Biological: Tozorakimab

INTERVENTIONS:
Biological: Tozorakimab — Tozorakimab will be administered as a single SC dose on Day 1.

SUMMARY:
The study will assess the relative bioavailability between two dosage forms of tozorakimab (test dosage form and reference dosage form) and to assess the pharmacokinetic (PK) profiles of both dosage forms.

DETAILED DESCRIPTION:
This is a phase I, randomised, open-label, single-dose, single-centre, parallel group study investigating the relative bioavailability of two dosage forms of tozorakimab (test dosage form and reference dosage form).

The study will comprise of:

1. A screening period of 28 days
2. A Treatment period of 1 day
3. Ambulatory visits on scheduled days

c. A final follow-up visit on Day 113 (Week 16)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants aged 18 to 55 years.
* All females must have a negative pregnancy test at the screening visit and on admission to the Clinical Unit.
* Females of childbearing potential must not be lactating and, if heterosexually active, must agree to use an approved method of highly effective contraception.
* Females of non-childbearing potential must be confirmed at the screening visit.
* Sexually active fertile male participants with partners of childbearing potential must adhere to the contraception methods.
* Have a body mass index (BMI) between 19 and 30 kg/m2 inclusive and weigh at least 55 kg and no more than 100 kg inclusive.
* Intact normal skin without potentially obscuring tattoos, scars, etc, at the injection site.

Exclusion Criteria:

* History of any clinically significant disease or disorder (including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment that is not stable in the opinion of the investigator).
* Any clinically significant abnormal findings in vital signs at the screening visit and/or admission (Day -1) to the Clinical Unit, as judged by the investigator.
* Any clinically significant abnormalities on 12-lead ECG at the screening visit and/or admission (Day -1) to the Clinical Unit, as judged by the investigator.
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the previous 6 months prior to the screening visit, as judged by the investigator.
* Any clinically important illness, medical/surgical procedure, or trauma within 8 weeks of the screening visit, or any planned inpatient surgery or hospitalisation during the study period.
* Malignancy, current or within the past 5 years, except for adequately treated non-invasive basal cell and squamous cell carcinoma of the skin and cervical carcinoma-in-situ treated with apparent success more than 1 year prior to enrolment. Suspected malignancy or undefined neoplasms.
* Suspicion of, or confirmed, ongoing SARS-CoV-2 infection.
* Any laboratory values with the following deviations at the screening visit or on admission (Day -1) to the Clinical Unit.
* Any clinically significant abnormal findings in physical examination at screening and/or admission (Day -1), which, in the opinion of the investigator, may put the participant at risk because of their participation in the study or may influence the results of the study, or the participant's ability to complete the entire duration of the study.
* History of known immunodeficiency disorder, including a positive test for Human immunodeficiency virus-1 (HIV-1) or HIV-2.
* History or treatment for hepatitis B or hepatitis C or any positive test result on screening for Hepatitis B surface antigen (HBsAg), anti- Hepatitis B core (HBc) antibodies, or anti-hepatitis C antibodies.
* Evidence of active or latent Tuberculosis (TB).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time 0 to infinity (AUCinf) | Day 1 (Pre-dose), Days 3, 4, 5, 7, 8, 9, 15, 29, 43, 57, 85 and 113 (Post-dose).
  To evaluate the relative bioavailability of two different dosage forms of tozorakimab (test and reference).
Area under the concentration-curve from time 0 to the last quantifiable concentration (AUClast) | Day 1 (Pre-dose), Days 3, 4, 5, 7, 8, 9, 15, 29, 43, 57, 85 and 113 (Post-dose).
  To evaluate the relative bioavailability of two different dosage forms of tozorakimab (test and reference).
Maximum observed drug concentration (Cmax) | Day 1 (Pre-dose), Days 3, 4, 5, 7, 8, 9, 15, 29, 43, 57, 85 and 113 (Post-dose).
  To evaluate the relative bioavailability of two different dosage forms of tozorakimab (test and reference).

SECONDARY OUTCOMES:
Time to reach peak or maximum observed concentration following tozorakimab administration (tmax) | Day 1 (Pre-dose), Days 3, 4, 5, 7, 8, 9, 15, 29, 43, 57, 85 and 113 (Post-dose).
  To examine the tmax of two different dosage forms of tozorakimab (test and reference).
Terminal elimination half-life (t1/2) | Day 1 (Pre-dose), Days 3, 4, 5, 7, 8, 9, 15, 29, 43, 57, 85 and 113 (Post-dose).
  To examine the t1/2 of two different dosage forms of tozorakimab (test and reference).
Terminal rate constant (λz) | Day 1 (Pre-dose), Days 3, 4, 5, 7, 8, 9, 15, 29, 43, 57, 85 and 113 (Post-dose).
  To examine the λz of of two different dosage forms of tozorakimab (test and reference).
Apparent total body clearance (CL/F) | Day 1 (Pre-dose), Days 3, 4, 5, 7, 8, 9, 15, 29, 43, 57, 85 and 113 (Post-dose).
  To examine the CL/F of two different dosage forms of tozorakimab (test and reference).
Apparent volume of distribution based on the terminal phase (Vz/F) | Day 1 (Pre-dose), Days 3, 4, 5, 7, 8, 9, 15, 29, 43, 57, 85 and 113 (Post-dose).
  To examine the Vz/F of two different dosage forms of tozorakimab (test and reference).
Number of participants with adverse events (AEs) | From screening (Day -28) to last follow-up visit (Day 113- approximately 21 weeks).
  To assess the safety and tolerability of a single dose of tozorakimab administered subcutaneously via two different dosage forms in healthy participants.
Number of participants with presence of Anti-Drug Anitbodies (ADAs) | Day 1 (Pre-dose), Days 29, 57 and 113 (Post-dose).
  To evaluate the immunogenicity of a single dose of tozorakimab administered subcutaneously via two different dosage forms in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/